CLINICAL TRIAL: NCT06445257
Title: A Prospective, Multicenter, Open-label, Single-arm Clinical Study Evaluating the Safety and Efficacy of ZRMT Regimen in the Treatment of Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of ZRMT Regimen in the Treatment of PCNSL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Collaborators: Affiliated Hospital of Nantong University (Other); The First People's Hospital of Changzhou (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2023-044-02
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — zanubrutinib; Rituximab; Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The ZRMT regimen is used to treat PCNSL (Experimental): zanubrutinib 160 mg BID orally rituximab: 375 mg/m2 intravenously on day 7, methotrexate: 3-3.5 g/m2 intravenously on day 1, and temozolomide 100 mg on days 1-5.
  Treatment will be given for 6-8 cycles, and patients who achieve a partial response (PR) or better can choose to undergo ASCT if they meet the transplantation criteria. After transplantation or for patients who do not undergo transplantation, zanubrutinib monotherapy maintenance treatment will be administered at a dose of 160 mg BID orally for 2 years or until disease progression, death, or intolerable adverse reactions.
  Interventions: Drug: zanubrutinib 160 mg BID orally

INTERVENTIONS:
Drug: zanubrutinib 160 mg BID orally — The ZRMT induction and maintenance regimen
  Other Names: rituximab: 375 mg/m2 intravenously on day 7; methotrexate: 3-3.5 g/m2 intravenously on day 1; temozolomide 100 mg on days 1-5

SUMMARY:
This study is a prospective, multicenter, open-label, single-arm clinical trial evaluating the safety and efficacy of the ZRMT (Zanubrutinib-Rituximab-Methotrexate-Temozolomide) regimen in the treatment of primary central nervous system lymphoma (PCNSL) with diffuse large B-cell lymphoma.

This study includes an induction phase for PCNSL ± ASCT and a sequential maintenance phase.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter, phase II clinical trial aimed at evaluating the safety, tolerability, and preliminary efficacy of ZRMT regimen ± ASCT followed by sequential zebutinib monotherapy as maintenance treatment for newly diagnosed PCNSL. A total of 30 subjects are planned to be enrolled.

Primary central nervous system lymphoma (PCNSL) accounts for only 1-2% of non-Hodgkin lymphoma (NHL) patients, with over 90% of PCNSL cases being diffuse large B-cell lymphoma. PCNSL is characterized by an aggressive clinical course and poor prognosis, with a 5-year overall survival (OS) rate of only 30.1% even with intensive chemotherapy and autologous stem cell transplantation as first-line consolidation. Additionally, the median age of onset for PCNSL is close to 70 years. Therefore, a low-toxicity and highly effective treatment regimen is crucial in the management of PCNSL. Currently, the standard treatment for PCNSL is combination chemotherapy based on high-dose methotrexate (HD-MTX), which has improved the survival of PCNSL patients compared to previous surgical resection or whole-brain radiation therapy. However, the efficacy of HD-MTX is not durable, with only 20% of patients achieving sustained remission after 2 years of HD-MTX monotherapy.

Young and healthy patients with PCNSL are recommended to undergo ASCT consolidation therapy in CR1 phase after intensified induction. However, approximately 25-35% of PCNSL patients are aged 70 or above, and these patients may not be suitable candidates for ASCT. Therefore, the treatment options for elderly and frail PCNSL patients still require further research.

Studies have shown that PCNSL is primarily of the ABC subtype of DLBCL. Whole exome sequencing has revealed that PCNSL patients typically have mutations in the MYD88 and CD79B genes, leading to the classification of PCNSL as the MCD subtype. Both of these genes are key molecules in the BCR signaling pathway. Mutations in MYD88 and CD79B ultimately lead to activation of NF-кB, promoting tumor cell proliferation and inhibiting apoptosis. The high frequency and functional activation of this pathway also provide new targets for treatment.The non-receptor tyrosine kinase Bruton tyrosine kinase (BTK) is a key molecule in the B-cell receptor (BCR) signaling pathway and is involved in the activation and survival of ABC subtype DLBCL cells. The BTK inhibitor Ibrutinib has shown promising anti-tumor activity in relapsed/refractory DLBCL, with higher response rates observed in ABC subtype patients compared to germinal center subtype patients (5% vs 37%, p=0.0106).

Zanbrutinib is a novel and potent covalent selective inhibitor of Bruton tyrosine kinase (BTK). Currently, the FDA has approved zanbrutinib for the treatment of relapsed/refractory chronic lymphocytic leukemia, mantle cell lymphoma, marginal zone lymphoma, and Waldenström macroglobulinemia, which are B-cell lymphomas. It is actively being studied and explored in other B-cell tumors, including diffuse large B-cell lymphoma, and promising efficacy and safety data are being reported gradually.In a multicenter, single-arm phase 2 study, 41 patients with relapsed/refractory DLBCL were treated with oral zanbrutinib at a dose of 160 mg twice daily until disease progression or intolerable toxicity. With a median follow-up of 6.8 months, the overall response rate (ORR) was 29.3%, with a complete response (CR) rate of 17.1%. The median duration of response (DOR), progression-free survival (PFS), and overall survival (OS) were 4.5, 2.8, and 8.4 months, respectively. This study preliminarily demonstrates the efficacy of zanbrutinib in central nervous system-involved DLBCL. Recent studies presented at ASH suggest that regimens containing BTK inhibitors show promising efficacy in first-line treatment of PCNSL, and the exploration of novel drug combinations with chemotherapy holds the potential to bring deeper and more durable remissions for PCNSL patients. However, further investigation is needed to determine the optimal drug combinations.

The main objective of this study is to evaluate the safety, tolerability, and preliminary efficacy of the ZRMT regimen in the treatment of newly diagnosed PCNSL. The secondary objective is to assess the preliminary efficacy of the ZRMT regimen ± ASCT followed by sequential maintenance therapy with zanubrutinib.After screening, eligible patients will receive zanubrutinib 160 mg BID orally, rituximab: 375 mg/m2 intravenously on day 7, methotrexate: 3-3.5 g/m2 intravenously on day 1, and temozolomide 100 mg on days 1-5. Treatment will be given for 6-8 cycles, and patients who achieve a partial response (PR) or better can choose to undergo ASCT if they meet the transplantation criteria. After transplantation or for patients who do not undergo transplantation, zanubrutinib monotherapy maintenance treatment will be administered at a dose of 160 mg BID orally for 2 years or until disease progression, death, or intolerable adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* According to the 2016 WHO classification of hematopoietic and lymphoid tissue tumors, the patient has been histopathologically diagnosed with primary central nervous system diffuse large B-cell lymphoma.
* Age ≥18 years and ≤75 years, any gender.
* Performance status score (ECOG): 0-1.
* Male participants and reproductive-age females must use contraception during the study and for 3 months after the last dose.
* Reproductive-age females must have a negative serum or urine pregnancy test at screening.
* Expected survival of more than 3 months.
* Laboratory tests must meet the following criteria:Hematology: Hemoglobin (Hb) ≥80 g/L, absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count (PLT) ≥75 × 109/L.Liver function: Serum total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤2.5 × ULN, alanine aminotransferase (ALT) ≤2.5 × ULN.Renal function: Creatinine clearance rate (Ccr) ≥50 mL/min.Coagulation function: International normalized ratio (INR) and prothrombin time (PT) ≤1.5 × ULN.Note: Patients who do not meet the above criteria may receive supportive treatment at the discretion of the investigator.
* The patient is aware of and voluntarily agrees to participate in the study and is able to comply with the scheduled visits and related procedures as specified in the protocol.

Exclusion Criteria:

* Patients who are determined by the investigator to be allergic, resistant, or intolerant to the drugs in the treatment regimen.
* Patients who have received any investigational drugs or radiation therapy within the past 4 weeks.
* Patients who have undergone major surgery within the past 4 weeks (excluding surgery related to the disease).
* Patients with severe infections within the past 4 weeks, as determined by the investigator, who are not suitable for treatment.
* Patients with a history of stroke or intracranial hemorrhage within the past 3 months, or active grade 3 or higher gastrointestinal bleeding.
* Patients who are pregnant or breastfeeding.
* Patients with impaired cardiac function or significant cardiac diseases, including but not limited to: a) myocardial infarction, congestive heart failure, or viral myocarditis within the past 6 months; b) symptomatic cardiac diseases requiring treatment intervention, such as unstable angina or arrhythmias; c) NYHA class II-IV heart function; d) echocardiographic ejection fraction (EF) below 50% or below the lower limit of the study center.
* Patients with a known history of human immunodeficiency virus (HIV) infection, primary immunodeficiency diseases, or active tuberculosis.
* Patients with poorly controlled hypertension or diabetes.
* Patients with active hepatitis B or hepatitis C infection (for HBsAg-positive or HBcAb-positive subjects, they can be included if HBV-DNA is not detected; for HCV antibody-positive subjects, they can be included if HCV-RNA is not detected).
* Patients with a history of malignant tumors that may affect the implementation of the trial protocol or result analysis (excluding cured basal cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast, localized gastric or intestinal mucosal carcinoma, and localized prostate cancer).
* Patients with active mental disorders, alcoholism, drug abuse, or substance abuse.
* Patients who are determined by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate，ORR | The period of 1 year from the start of treatment.
  Refers to the proportion of patients whose tumor volume has decreased to a predetermined value and can be maintained for a minimum duration requirement
Complete response，CR | The period of 1 year from the start of treatment
  refers to the time from the first assessment of CR or PR to the first assessment of PD or death for any reason
Duration of response,DOR | The period of 1 year from the start of treatment
  refers to the time from the first assessment of CR or PR to the first assessment of PD or death for any reason
1 Year-Overall survival,1y-OS | The period of 1 year from the start of treatment
  refers to the proportion of patients who have not died within 1 year after the start of the first treatment.
Progression-Free Survival,PFS | The period of 1 year from the start of treatment
  refers to the proportion of patients who have not experienced disease progression or death within 1 year after the start of the first treatment
Overall survival, OS | The period of 1 year from the start of treatment
  refers to the time from the start of the first treatment to death (for any reason)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University（Huai'an First People's Hospital）, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No